CLINICAL TRIAL: NCT02277262
Title: PROPHYlactic Implantation of BIOlogic Mesh in Peritonitis (PROPHYBIOM)
Acronym: PROPHYBIOM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: A.O. Ospedale Papa Giovanni XXIII (Other)
Responsible Party: Principal Investigator, Federico Coccolini, General Surgeon, A.O. Ospedale Papa Giovanni XXIII
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 154-14
Record Dates: First submitted 2014-10-14; First posted 2014-10-28 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Incisional Hernia
Keywords: peritonitis patients
MeSH Terms: conditions — Incisional Hernia

ARMS (2):
- Treatment arm (Experimental): Patients randomized to this arm will be operated for the primary disease and at the end of the intervention the laparotomy will be closed reinforcing the suture with a swine dermis biological prosthesis positioned sublay
  Interventions: Device: Biological swine dermis not cross-linked prosthesis positioning in incisional hernia prevention
- Control arm (Active Comparator): Patients randomized to this arm will be operated for the primary disease and at the end of the intervention the laparotomy will be closed by emi-continuous monofilament sutures with an intermediate-reabsorbable-time suture
  Interventions: Procedure: Direct suture of the anterior abdominal wall fascia

INTERVENTIONS:
Device: Biological swine dermis not cross-linked prosthesis positioning in incisional hernia prevention — The mesh placement will be preceded by the plane preparation. The subcutaneous tissue will be dissociated from the anterior rectum-muscles fascia. The retro-muscular rectum muscles plane will be dissected preparing a 5-6 cm pouch necessary to the prosthesis positioning. The mesh will be fixed with at least 8 long-lasting absorbable transfix stitched. The prosthesis will be placed with at least a 5 cm overlap. If the peritoneal plane can be sutured a Jackson-Pratt 10 suction drain will be placed under the prosthesis. A Jackson-Pratt 10 suction drain will always be placed over the prosthesis. Anterior rectum fascia will be closed by emi-continuous monofilament suture with an intermediate-reabsorbable-time suture. Another Jackson-Pratt 10 suction drain will be placed over the anterior fascia if the subcutaneous tissue is thick. No subcutaneous suture will be performed. Skin stapler or interrupted stitches will be used to close the skin plane.
  Other Names: Biological swine dermis not-cross-linked prosthesis positioning
  Arms: Treatment arm
Procedure: Direct suture of the anterior abdominal wall fascia — Anterior rectum fascia will be closed by emi-continuous monofilament suture with an intermediate-reabsorbable-time suture. No subcutaneous suture will be performed. Skin stapler or interrupted stitches will be used to close the skin plane.
  Arms: Control arm

SUMMARY:
To evaluate the efficacy of the use of swine dermal collagen prosthesis implanted preperitoneally as a prophylactic procedure against incisional hernia in patients operated in urgency/emergency setting in contaminated/infected fields with peritonitis. The aim of the study is to reduce the incidence of incisional hernia from 50% to 20%.

ELIGIBILITY:
Inclusion Criteria:

* • Patients aged > 18 years old

  * Clinical and/or laboratory and/or radiological evidence/signs of peritonitis of any origin (peritoneal reactivity, positive Blumberg sign, fever, free air/fluid in abdominal cavity, leucocytosis, increased CRP (C-reactive protein, lactic dehydrogenase (LDH), tachycardia, tachypnea, clinical or radiological evidence/suspect of bowel ischemia)
  * Eventual strong suspect of possible bacterial translocation (reduction of the natural intestinal barrier against bacterial translocation, i.e. bowel ischemia, bowel overdistension, intestinal occlusion, etc.)
  * Surgical indication for midline laparotomy independently from eventual previous laparotomies
  * Informed consent

Exclusion Criteria:

* • Patients aged < 18 years old

  * Informed consent refusal
  * No Clinical and/or laboratory and/or radiological evidence/signs of peritonitis of any origin.
  * Surgical indication for laparotomies other than midline one
  * Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Incisional hernia rate | 3 months
Incisional hernia rate | 6 months
Incisional hernia rate | 12 months
Incisional hernia rate | 24 months

SECONDARY OUTCOMES:
Morbidity | 0 months
Morbidity | 3 months
Morbidity | 6 months
Morbidity | 12 months
Morbidity | 24 months
Length of surgery | Day 0
Time to drain removal | participants will be followed for the duration of hospital stay, an expected average of 1-2 weeks
Length of stay in hospital | At the discharge, an expected average of 1-2 weeks after the intervention
Mortality | 0 months
Mortality | 3 months
Mortality | 6 months
Mortality | 12 months
Mortality | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Papa Giovanni XXIII hospital, Bergamo, Italy